CLINICAL TRIAL: NCT01222611
Title: Randomized, Controlled, Open Label, Pilot Study to Evaluate Fosamprenavir Activity on Genotype 1 Hepatitis C Virus (HCV) Infection Evolution in Human Immunodeficiency Virus (HIV) Co-infected Subjects With Antiretroviral Treatment Including Fosamprenavir
Brief Title: HCV Evolution in HIV/HCV (Genotype 1) Coinfected Patients Treated With Fosamprenavir
Acronym: FOSTER-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 6710; 2010-023503-10 (EudraCT Number)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-09

CONDITIONS: Chronic HIV Infection; HCV Coinfection
Keywords: HIV; HCV; HIV/HCV; Coinfection; Fosamprenavir
MeSH Terms: conditions — Coinfection | interventions — fosamprenavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard HAART (No Intervention): ART with 3 drugs including 2 NRTIs plus a ritonavir boosted PI (different to FPV) or a NNRTI
- HAART inlcuding Fos APV/r (Experimental): ART with 3 drugs including 2 NRTIs plus ritonavir boosted fosamprenavir
  Interventions: Drug: Fosamprenavir

INTERVENTIONS:
Drug: Fosamprenavir — HAART including fosamprenavir boosted with ritonavir
  Other Names: Telzir(r)
  Arms: HAART inlcuding Fos APV/r

SUMMARY:
This study examines the impact of fosamprenavir as part of an ART on virological, immunological and clinical parameters of genotype 1 HCV infection in HIV co-infected subjects. Fosamprenavir could have a direct or immune-mediated activity against HCV. If this is shown to be true, changes in HCV viral load or biological characteristics could be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yo
* HIV/HCV co-infected patients with HCV detectable viremia in 2 determinations separated at least by 6 months.
* HCV genotype 1
* Currently receiving ART including 2NRTI+1 PI/r (excluding FPV) or 1 NNRTI, without changes in the last 6 months
* HIV RNA < 50 copies/mL for the last 6 months

Exclusion Criteria:

* Previous anti HCV treatment
* Foreseeable HCV treatment in the next 12 months
* Acute HCV infection
* Active opportunistic infection
* HIV with FPV resistance mutations
* Current or previous treatment with FPV
* Chronic hepatitis B
* Current alcohol consumption greater than 20 g per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
HCV Viral load and changes in HCV protease gene | 48 weeks
  Undetectable HCV viral load. It will be considered that one patient achieves this endpoint if he/she has an undetectable HCV viral load (<30 copies/mL) at any time during the study. If a patient shows undetectable HCV viral load and afterwards shows a detectable load, it will be considered that this patient achieved this endpoint.
  Changes in the HCV protease gen. Any change from baseline in the protease catalytic domain, analysed by population sequencing of the catalytic domain of the HCV protease.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gonzalez, MD, Principal Investigator — Hospital La Paz, Madrid (Spain)
Locations (6):
- Spain (6):
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid